CLINICAL TRIAL: NCT03986151
Title: Anatomical sNuffbox for Coronary anGiography and IntervEntions
Acronym: ANGIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Grigorios Tsigkas, Cardiology consultant, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11994/6-5-2019
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Vascular Access Complication
Keywords: coronary angiography; radial access; distal radial access; anatomical snuffbox; radial artery occlusion
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radial access (Active Comparator)
  Interventions: Procedure: Coronary angiography +/- percutaneous coronary intervention
- Distal radial access (Experimental)
  Interventions: Procedure: Coronary angiography +/- percutaneous coronary intervention

INTERVENTIONS:
Procedure: Coronary angiography +/- percutaneous coronary intervention — Comparison of the conventional radial approach with the distal radial approach (anatomical snuffbox)

SUMMARY:
This randomized, single-center, prospective study seeks to compare the conventional radial approach with the recently described distal radial approach (anatomical snuffbox) concerning the patency of the radial artery in patients subjected to coronary angiography or percutaneous coronary intervention.

DETAILED DESCRIPTION:
Transradial approach has become the standard approach for coronary angiography (CAG) and percutaneous coronary intervention (PCI). The current ESC/EACTS guidelines of myocardial revascularization support using radial approach (RA) rather than femoral approach (FA) if the operators are experts for RA. Recently, an alternative transradial access has been suggested at the anatomical snuffbox, with potential additional benefits including a reduction in radial artery occlusion rate (which allows reintervention through the same access site and potential use as a graft), a decrease in other local vascular complications, shorter hemostasis duration, patients' intra and post procedural comfort and shorter recovery time. However, the feasibility of PCI via snuffbox approach is still concerned due to the lack of data. Therefore, the aim of the study is to compare the two approaches concerning the patency of the radial artery ≥30 days after the intervention with Doppler in a randomized way. Due to the anastomosis of the distal radial artery with the superficial palmar arch, even in case of total radial artery occlusion within the anatomical snuffbox, the antegrade blood flow may be preserved and, therefore, decreased incidents of radial artery occlusion are expected in the right distal radial artery approach group. The mean diameter of radial artery at the anatomical snuffbox is 2.4 mm, whereas the mean diameter of the radial artery at the forearm is 2.7 mm, and this could potentially contribute to shorter hemostasis duration.

ELIGIBILITY:
Inclusion Criteria:

* Indication for coronary angiography
* Informed consent

Exclusion Criteria:

* Non palpable right radial artery
* Prior complicated right transradial intervention (radial artery dissection, perforation, occlusion)
* Prior CABG
* STEMI
* Hemodynamic instability
* Anatomical restrictions (fistula, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Rate of right radial artery occlusion | ≥30 days after CAG or PCI

SECONDARY OUTCOMES:
Rate of successful insertion of the sheath | Immediately post-procedurally
Duration of sheath insertion procedure | Immediately post-procedurally
Rate of successful completion of coronary angiography | Immediately post-procedurally
Rate of successful completion of percutaneous coronary intervention | Immediately post-procedurally
Total Contrast volume | Immediately post-procedurally
Total Fluoroscopy time | Immediately post-procedurally
Total Radiation Dose | Immediately post-procedurally
Total Procedure Time | Immediately post-procedurally
Time required for hemostasis | 1-6 hours
Postprocedural Hematoma (modified EASY class) | 3 hours
Rate of distal radial artery occlusion | ≥30 days after CAG or PCI
Pain associated with the procedure: Pain scale 0-10 | 1 hour
  Pain scale 0-10. A visual anlog pain scale 0-10 will be shown to the patient post-precedurally. 0=no pain, 10=worst pain. Patient will be asked to report the severity of the pain associated with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Tsigkas, MD, Phd, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Yes